CLINICAL TRIAL: NCT01847638
Title: Clinical Outcomes of Prolensa (Bromfenac Ophthalmic Solution) 0.07% QD vs. Ilevro (Nepafenac Ophthalmic Suspension) 0.3% QD for Treatment of Ocular Inflammation Associated With Cataract Surgery
Brief Title: Prolensa (Bromfenac) 0.07% QD vs. Ilevro (Nepafenac) 0.3% QD for Treatment of Ocular Inflammation Post Cataract Surgery
Acronym: QD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melissa Toyos (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Melissa Toyos, Principal Investigator, Toyos Clinic
Organization: Toyos Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMT-2013
Record Dates: First submitted 2013-04-16; First posted 2013-05-07 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Cataract; Retinal Edema; Inflammation
Keywords: Retinal edema; Cataract; inflammation
MeSH Terms: conditions — Cataract; Papilledema; Inflammation | interventions — bromfenac; nepafenac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolensa (bromfenac 0.07%) (Active Comparator): Subjects will instill one drop Prolensa (bromfenac 0.07%) into the study (operative) eye once daily for a maximum of 25 days. Dosing will begin three days prior to surgery (Day 3), continue on the day of surgery and for 21 days after surgery.
  Interventions: Drug: Prolensa (bromfenac 0.07%)
- Ilevro (nepafenac 0.3%) (Active Comparator): Subjects will instill one drop into the study (operative) eye once daily for a maximum of 25 days. Dosing will begin three days prior to surgery (Day 3), continue on the day of surgery and for 21 days after surgery.
  Interventions: Drug: Ilevro (nepafenac 0.3%)

INTERVENTIONS:
Drug: Prolensa (bromfenac 0.07%) — Comparison of Prolensa (bromfenac ophthalmic solution) 0.07% QD vs. Ilevro (nepafenac ophthalmic suspension) 0.3% QD for Treatment of Ocular Inflammation Associated with Cataract Surgery
  Other Names: bromfenac ophthalmic solution 0.07%
  Arms: Prolensa (bromfenac 0.07%)
Drug: Ilevro (nepafenac 0.3%) — Comparison of Prolensa (bromfenac ophthalmic solution) 0.07% QD vs. Ilevro (nepafenac ophthalmic suspension) 0.3% QD for Treatment of Ocular Inflammation Associated with Cataract Surgery
  Other Names: nepafenac ophthalmic suspension 0.3%
  Arms: Ilevro (nepafenac 0.3%)

SUMMARY:
To investigate inflammation, visual acuity and macular thickness after treatment with Prolensa vs Ilevro after cataract surgery.

DETAILED DESCRIPTION:
To investigate the clinical outcomes for inflammation, visual acuity and macular thickness after treatment with Prolensa (bromfenac ophthalmic solution) 0.07% QD in subjects who have undergone cataract extraction with posterior chamber intraocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female at least 18 years of age who require cataract surgery and no other surgical procedures during the cataract surgery.
* Agree not to have any other ocular surgical procedures in the study or fellow (non study) eye within 15 days prior to the initiation of dosing with the test article or throughout the duration of the study.
* Have a Best Corrected Visual Acuity of 20/200 or better in either eye.
* Are able to self administer test article (or have a caregiver available to instill all doses of test article).

Exclusion Criteria:

* Have known hypersensitivity to bromfenac, nepafenac, loteprednol or any component of the test article (including "procedural" medications such as anesthetic and/or fluorescein drops, dilating drops, etc.).
* Have a known hypersensitivity to salicylates (i.e., aspirin) or NSAIDs (nonsteroidal antiinflammatory drug).
* Have intraocular inflammation (i.e., cells or flare in the anterior chamber as measured on slit lamp examination) in study eye at screening visit.
* Have a known blood dyscrasia or bone marrow suppression, a diagnosis of uncontrolled/unstable peptic ulcer disease, inflammatory bowel disease, or ulcerative colitis, or any uncontrolled/unstable pulmonary, cardiac, vascular, autoimmune, hepatic, renal, or central nervous system disease.
* Have used ocular, topical, or systemic NSAIDs or ocular, topical, or systemic gentamicin, or cyclosporine ophthalmic emulsion within 7 days prior to initiation of dosing with the test article or throughout the duration of study,with exception of allowing patients on a stable dose of aspirin 81 mg daily or less.
* Have used ocular prostaglandins within 30 days prior to initiation of dosing with test article or throughout the duration of study.
* Have active corneal pathology noted in the study eye at screening visit. Active corneal pathology is defined as corneal pathology that is non stable, or greater than mild, or will compromise assessment of the safety or efficacy of treatment. Superficial punctate keratitis in study eye.
* Have any extraocular/intraocular inflammation in the study eye at screening visit (blepharitis allowed if mild only, and no concurrent conjunctivitis or lid erythema/edema) or ongoing, unresolved uveitis.
* Have used topical, ocular, inhaled or systemic steroids within 14 days prior to screening.
* Have had radial keratotomy, corneal transplant, or corneal refractive surgery in the study eye within the last two years.
* Have a history of abuse of alcohol/drugs within six months prior to the screening visit.
* Are pregnant or nursing/lactating.
* Have participated in any other study of an investigational drug or device within 30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2018-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Toyos, MD, Principal Investigator — Toyos Clinic
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Toyos MM. Comparison of Once-Daily Bromfenac 0.07% Versus Once-Daily Nepafenac 0.3% in Patients Undergoing Phacoemulsification. Ophthalmol Ther. 2019 Jun;8(2):261-270. doi: 10.1007/s40123-019-0174-x. Epub 2019 Mar 13. PMID 30868419

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prolensa (Bromfenac 0.07%) | Ilevro (Nepafenac 0.3%)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolensa (Bromfenac 0.07%) | Ilevro (Nepafenac 0.3%) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 20 | 32
  >=65 years | 13 | 5 | 18
Age, Continuous [Mean (Full Range); unit: years] | 68.3 [53 to 85] | 66.9 [48 to 87] | 67.6 [48 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Treatment of Inflammation Associated With Cataract Surgery
Description: Units on a scale. Biomicroscopy with slit lamp beam of 0.3 mm in width and 1.0 mm in height will be used to determine anterior cell and flare scores at each study visit by counting each individual white blood cell present and grading the flare (measure of protein and marker of inflammation in aqueous fluid). The sum of the severity of cell count and the flare grade will be called the Summed Ocular Inflammation Score (SOIS) and measured at each time point. The scale is 0-4 range for both values cells counted and flare where 0=no cell and 0=complete abscence of flare; 0.5 = 1-5 cells (trace) and 0= no flare; 1=6-15 cells and 1=very slight (barely detectable ) flare, 2=16-25 cells and 2=moderate flare (iris and lens clear), 3=26-30 cells and 3 =marked (iris and lens hazy) and 4=>
Time Frame: change from baseline to final at post op 42 days +/-7 days
Population: patients undergoing uncomplicated cataract surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolensa (Bromfenac 0.07%) | Ilevro (Nepafenac 0.3%)
Number analyzed (Participants) | 25 | 25
units on a scale | 0.01 (.3) | 0.01 (.4)

2. Secondary Outcome: Visual Acuity
Description: ETDRS log MAR Visual Acuity from baseline to final postoperative visit. The change was calculated as the difference of the value at the later time point minus the value at the earlier time point. The scale runs from -0.30 (corresponding to 20/10) or better visual acuity to 1(20/200) or worse visual acuity with the smaller or more negative numbers indicating better visual acuity outcomes and larger numbers indicating worsened visual acuity outcomes.
Time Frame: baseline score to final postoperative visit at 42 days +/-7 days
Population: patients undergoing uncomplicated cataract surgery
Measure: Mean (Standard Deviation); unit: logMar
Arm/Group | Prolensa (Bromfenac 0.07%) | Ilevro (Nepafenac 0.3%)
Number analyzed (Participants) | 25 | 25
logMar | .19 (.2) | .21 (.25)

3. Other Pre Specified Outcome: Retinal Thickness
Description: Change in Retinal Thickness from baseline to final postoperative visit as measured by an SD-OCT
Time Frame: change from baseline to final postoperative visit at 42 days +/- 7 days
Population: Patients undergoing uncomplicated phacoemulsification with lens implantation at a single center by a single surgeon.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Prolensa (Bromfenac 0.07%) | Ilevro (Nepafenac 0.3%)
Number analyzed (Participants) | 25 | 25
microns | 276 (1.26) | 279 (2.1)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Prolensa (Bromfenac 0.07%) | Ilevro (Nepafenac 0.3%)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolensa (Bromfenac 0.07%) (N=25) | Ilevro (Nepafenac 0.3%) (N=25)
iritis (Eye disorders) | 1 (1) | 0 (0) — iritis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No